CLINICAL TRIAL: NCT00424164
Title: Pharmacokinetics Study of Combined Treatment Lapatinib and Tamoxifen in Advanced/Metastatic Breast Cancer
Brief Title: Lapatinib and Tamoxifen in Treating Patients With Advanced or Metastatic Breast Cancer
Acronym: LAPATAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10053; 2005-005196-14 (EudraCT Number)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Lapatinib; Tamoxifen

ARMS (2):
- Tamoxifen-lapatinib (Experimental): Tamoxifen alone at cycle 1 and as of cycle 2 in combination with Lapatinib.
  Interventions: Drug: lapatinib ditosylate; Drug: tamoxifen citrate; Other: pharmacological study
- Lapatinib-tamoxifen (Experimental): Lapatinib will be given alone for 2 weeks during cycle 1. As of cycle 2, you will receive the combined treatment Lapatinib and Tamoxifen
  Interventions: Drug: lapatinib ditosylate; Drug: tamoxifen citrate; Other: pharmacological study

INTERVENTIONS:
Drug: lapatinib ditosylate
Drug: tamoxifen citrate
Other: pharmacological study

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving lapatinib together with tamoxifen may be an effective treatment for breast cancer.

PURPOSE: This randomized phase I trial is studying the side effects of lapatinib and tamoxifen in treating patients with advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacokinetics of lapatinib ditosylate and tamoxifen citrate in patients with advanced or metastatic breast cancer.

Secondary

* Assess the safety of this regimen in these patients.
* Determine any relationship between drug exposure and adverse events or biological modifications of this regimen in these patients.
* Assess the antitumor activity of this regimen in patients with measurable disease.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen citrate on days 1-28 of course 1. In all subsequent courses, patients receive oral tamoxifen citrate and oral lapatinib ditosylate on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral lapatinib ditosylate on days 1-14 of course 1. In all subsequent courses, patients receive oral lapatinib ditosylate and oral tamoxifen citrate on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

In both treatment arms, blood is collected periodically during courses 1 and 2 for pharmacokinetic studies.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic breast cancer

  * Progressive disease after aromatase inhibitor therapy
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive tumor
* Patients with stable brain metastases (i.e., no neurological symptoms and no corticosteroid treatment) are eligible

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* AST and/or ALT < 3 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* Bilirubin < 1.5 times ULN
* Clinically normal cardiac function (i.e., LVEF normal by MUGA or ECHO)
* No current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic live disease)
* No ischemic heart disease within the past 6 months
* Normal 12-lead ECG
* No active or uncontrolled infections
* No serious illnesses or medical conditions, including any of the following:

  * Hypercalcemia
  * Malabsorption syndrome
  * Chronic alcohol abuse
  * Hepatitis
  * HIV
  * Cirrhosis
* Able to swallow and retain oral medication
* No psychological, familial, sociological, or geographical condition potentially hampering study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 days since prior and no concurrent inducers or inhibitors of CYP3A4, including any of the following:

  * Rifabutin
  * Clarithromycin
  * Cyclosporine
  * Voriconazole
  * Fluoxetine
  * Paroxetine
  * Midazolam
  * Isoniazid
  * Dihydralazine
  * Digitoxin
  * Coumadin
  * Phenytoin
  * Verapamil
  * Diltiazem
  * Herbal constituents (e.g., bergamottin and glabridin)
* At least 2 weeks since prior aromatase inhibitor

  * Aromatase inhibitors in the adjuvant and/or metastatic setting allowed
* At least 1 year since prior tamoxifen citrate
* No other concurrent anticancer therapy or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2010-05-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of lapatinib ditosylate and tamoxifen citrate alone and in combination | maximum 24h after the dose administered on Day 28

SECONDARY OUTCOMES:
Safety | until disease progression or until the start of another treatment (average 2 months)
Relationship between drug exposure and adverse events or biological modifications | until disease progression or until the start of another treatment (average 2 months)
Response in patients with measurable disease | until disease progression or until the start of another treatment (average 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (1):
- Centre Regional Rene Gauducheau, Dijon, France

REFERENCES:
- [Derived] Fumoleau P, Koch KM, Brain E, Lokiec F, Rezai K, Awada A, Hayward L, Werutsky G, Bogaerts J, Marreaud S, Cardoso F. A phase I pharmacokinetics study of lapatinib and tamoxifen in metastatic breast cancer (EORTC 10053 Lapatam study). Breast. 2014 Oct;23(5):663-9. doi: 10.1016/j.breast.2014.07.003. Epub 2014 Jul 24. PMID 25065668